CLINICAL TRIAL: NCT03082131
Title: Resistant Starch Wheat for Improved Metabolic Health: A Proof of Concept Study in Human Subjects
Brief Title: Resistant Starch Wheat for Improved Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 984621-1
Record Dates: First submitted 2017-03-10; First posted 2017-03-17 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Gut Microbiota; Metabolism; Metabolic Health
Keywords: Gut Microbiota; Glycemic Response; Resistant Starch; Fiber

STUDY DESIGN:
Intervention Model Description: Randomized, cross-over design consisting of two 1-week dietary intervention periods as well as a 2-week washout period in between
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be blinded to the type of product (i.e. RS wheat or Regular Wheat) the subjects are consuming during each arm of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Order of treatments:
  A. Resistant Starch Wheat B. Regular Wheat
  Interventions: Dietary Supplement: Resistant Starch Wheat
- Group 2 (Experimental): Order of treatments:
  A. Regular Wheat B. Resistant Starch Wheat
  Interventions: Dietary Supplement: Resistant Starch Wheat

INTERVENTIONS:
Dietary Supplement: Resistant Starch Wheat — The investigators will be testing high amylose wheat varieties developed by Arcadia Biosciences that have high levels of RS in the endosperm, the source of refined flour. Compared to regular wheat varieties with RS levels of less than 1%, Arcadia's wheat varieties contain between 16% and 34% RS.

SUMMARY:
The objective of this study is to determine the effect of wheat enriched in resistant starch (RS) on the generation of fermentation products by the lower gut microbes, the fecal microbiota profile, intestinal metabolites, and the glycemic response to a test meal compared to regular wheat.

DETAILED DESCRIPTION:
Resistant starch (RS) is a type of dietary fiber that provides fermentable carbohydrate (FC) in the lower bowel yielding positive effects on postprandial glycemia and weight management as well as digestive tract health. RS is defined as the portion of starch resistant to digestion by amylases, allowing it to reach the distal intestine where it can be fermented by the resident intestinal microbiota. A limited number of human studies using RS from high amylose corn have demonstrated that RS increases synthesis of gut peptides that improve glucose homeostasis and insulin secretion. Based on these studies, the FDA has recently approved the following health claims for resistant starch derived from corn (RS2): lowering of blood glucose, blood cholesterol, and blood pressure; increased mineral absorption; improved laxation; and reduced energy intake. The purpose in the proposed "proof of concept" study here is to show that RS provided in the form of wheat flour products has similar beneficial effects. The investigators aim to further explore the effect of RS on the gut microbiota. The intestinal microbiome is comprised of over one trillion bacterial cells comprised of approximately one thousand species that perform diverse functions ranging from energy harvest, angiogenesis, immunomodulation, and regulation of mood and behavior. Some of the major products of bacterial metabolism include acetate, propionate, and butyrate, the major short chain fatty acids (SCFA). These bioactive fermentation products have been associated with improved glucose homeostasis, attributed, in part, by their interactions with receptors on intestinal cells to augment secretion of glucagon-like peptide-1 (GLP-1), an incretin hormone known to stimulate insulin secretion.

This study is a randomized, cross-over design consisting of two 1-week dietary intervention periods as well as a 2-week washout period in between. Subjects will be randomly assigned to receive either RS wheat first or regular wheat first, then will be crossed over to the opposite treatment following a 2-week washout period. Wheat products made from RS wheat and regular wheat will be provided and the volunteers will be instructed to incorporate the products into their usual diet for 7 days. This study will probe the associations between the gut microbiota profiles, fermentation of RS wheat, microbial-mediated alterations in bile acids, and glycemia. The investigators will measure these effects in healthy, middle-aged humans using an interdisciplinary approach that integrates nutrition, microbiology, intestinal physiology, and analytical chemistry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults. Healthy means that the candidate reports that s/he feels well and can perform normal activities.

Exclusion Criteria:

* BMI <18.5 and >39.9 kg/m2
* Presence of of untreated or uncontrolled metabolic diseases
* Presence of gastrointestinal disorders that could interfere with the study outcome (i.e. Crohn's disease, Irritable bowel syndrome, Colitis)
* Use of oral antibiotics within the past 3 months
* Presence of cancer or other serious chronic disease by self report
* Current use of prescribed or over the counter weight loss medications
* Pregnant
* Lactating
* Current use of tobacco
* Dietary restrictions that would interfere with consuming the intervention foods

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Changes in Gut Microbiota Composition | Days 1, 7, 22, and 29
  Gut microbiota community composition will be determined by 16S ribosomal ribonucleic acid (rRNA) gene sequencing from stool samples

SECONDARY OUTCOMES:
Changes in Glucose Metabolism | 0, 1, 2, and 3 hours postprandial
  Fasting and postprandial measures of blood glucose, insulin, GLP-1
Changes in Gut Microbiota Metabolism | 0, 0.5, 1, 1.5, 2, 2.5, 3 hours postprandial
  Fasting and postprandial measures of hydrogen and methane in breath
Changes in Gut Microbiota Metabolism | 0, 1, 2, and 3 hours postprandial
  Fasting and postprandial measures of SCFA and bile acids in plasma
Evaluation of Consumer Acceptance | Days 8 and 30
  Participant-reported liking and taste
Dietary Intake | Days 3, 5, 8, 25, 27, and 30
  24-hour dietary recalls

CONTACTS AND LOCATIONS:
Locations (1):
- Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No